CLINICAL TRIAL: NCT03358329
Title: The ENCORE Study: Safety Evaluation of Repeat Placement of the Corticosteroid-Releasing S8 Sinus Implant in Chronic Sinusitis Patients With Nasal Polyps
Brief Title: Safety Evaluation of Repeat Placement of the S8 Sinus Implant in Chronic Sinusitis Patients With Nasal Polyps (ENCORE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P500-0717
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Chronic Sinusitis; Nasal Polyposis
Keywords: corticosteroid; implant
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S8 Sinus Implant (Experimental): corticosteroid-eluting sinus implant containing 1350 mcg of mometasone furoate (MF)
  Interventions: Combination Product: S8 Sinus Implant

INTERVENTIONS:
Combination Product: S8 Sinus Implant — In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses

SUMMARY:
The ENCORE Study is designed to evaluate the repeat administration of the S8 Sinus Implant in chronic sinusitis (CS) patients with recurrent nasal polyps.

DETAILED DESCRIPTION:
The ENCORE Study is a prospective open-label, non-randomized, multicenter study in CS patients who had undergone prior endoscopic sinus surgery (ESS) including bilateral total ethmoidectomy and present with bilateral ethmoid polyposis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent using a form approved by the reviewing institutional review board (IRB) and sponsor.
2. Patient is ≥ 18 years of age.
3. Patient is willing and able to comply with protocol requirements.
4. Patient has a confirmed diagnosis of CS with nasal polyps, as defined in the 2016 "International Consensus Statement on Allergy and Rhinology".
5. Patient has undergone prior ESS including bilateral total ethmoidectomy at least 90 days prior to screening.
6. Patient has evidence of bilateral ethmoid sinus obstruction due to polyposis warranting intervention (polyp grade ≥ 2 on each side).
7. Patient is able to tolerate daily use of Mometasone Furoate Nasal Spray (MFNS).
8. Patient is able to tolerate topical/local anesthesia.
9. In the opinion of the investigator, patient's ethmoid sinus anatomy is amenable to in-office bilateral placement of the S8 Sinus Implant (i.e., able to pass into the middle meatus on both sides the S8 Sinus Implant with 20 mm in nominal length and 7 mm in compressed diameter).
10. Female patients of reproductive potential must not be pregnant or nursing and must agree to not become pregnant during their participation in the study.
11. Female patients of childbearing potential must agree to use consistent and acceptable method(s) of birth control during their participation in the study.

Exclusion Criteria:

1. Patient has extensive ethmoid sinus polyp grade (grade 4 on at least one side).
2. Patient has extensive adhesions/synechiae (grade 3 or 4).
3. Patient has used parenteral and injected steroids (e.g., Kenalog injection) during 30 days prior to the baseline procedure.
4. Patient has used oral steroids, budesonide or other sinus steroid irrigations/rinses, nebulized steroids administered nasally or budesonide drops during 14 days prior to the baseline procedure.
5. Patient has oral-steroid dependent condition such as chronic obstructive pulmonary disease (COPD) or asthma.
6. Patient has known history of allergy or intolerance to corticosteroids or mometasone furoate.
7. Patient has used monoclonal antibodies for asthma, allergies or nasal polyps (e.g., Dupixent, Nucala, Xolair) during 30 days prior to the baseline procedure.
8. Patient requires monoclonal antibodies for asthma, allergies or nasal polyps during the duration of the study.
9. Patient has presence of physical obstruction that would preclude access and placement of the S8 Sinus Implant in the middle meatus (e.g., severe septal deviation, septal spur, very small middle meatus, total obstruction of the sinonasal passage with severe adhesion, scarring, polypoid edema or polyps).
10. Patient has known history of human immunodeficiency virus (HIV) or immunoglobulin G or A subclass deficiency.
11. Patient has clinical evidence of acute sinusitis (AS), as defined in the 2016 "International Consensus Statement on Allergy and Rhinology".
12. Patient has clinical evidence or suspicion of invasive fungal sinusitis (e.g., bone erosion on prior computed tomography (CT) scan, necrotic sinus tissue).
13. Patient has evidence of severe concomitant disease or condition expected to compromise survival or ability to complete assessments during the 365-day study follow-up period (e.g., cancer).
14. Patient is currently participating in another clinical study.
15. Patient has previously undergone ESS and experienced a cerebrospinal fluid (CSF) leak or has residual compromised vision as a result of a complication in a prior ESS procedure.
16. Patient has known dehiscence of the lamina papyracea.
17. Patient has evidence of active tuberculosis or active viral illness (e.g., ocular herpes simplex, chickenpox, measles).
18. Patient has known history or diagnosis of glaucoma or ocular hypertension (prior ocular exam with intraocular pressure of >21 mmHg and pressure lowering medication given) or posterior subcapsular cataract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Manes, MD, Principal Investigator — Yale University
Locations (9):
- United States (9):
  - Sacramento ENT, Sacramento, California
  - Yale University School of Medicine, New Haven, Connecticut
  - DuPage Medical Group, Naperville, Illinois
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Associated Surgical Specialists, Covington, Louisiana
  - BreatheAmerica of Albuquerque, Albuquerque, New Mexico
  - Madison ENT, New York, New York
  - Charlotte Eye, Ear, Nose and Throat Associates, Concord, North Carolina
  - Bridgerland Clinical Research, North Logan, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 10 sites across the US between November 2017 and January 2018.
Groups:
- S8 Sinus Implant: Corticosteroid-eluting Sinus Implant with 1350 mcg of MF
  Mometasone furoate nasal spray (200 mcg) once daily
Period: Overall Study
Arm/Group | S8 Sinus Implant
Started | 50
Completed | 46
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | S8 Sinus Implant
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46
  Black or African American | 2
  Asian | 1
  Other | 1
SNOT-22 [Mean (Standard Deviation); unit: units on a scale] — Sino-Nasal Outcomes Test (SNOT-22) is a validated disease-specific symptom-scoring instrument consisting of 22 questions, each scored on a 6-point scale of 0 (no problem) to 5 (probably as bad as it can be) based on the subject's recollection of symptoms over the past 2 weeks. The total score ranges from 0 to 110, with a higher score reflecting greater symptom burden. Negative values for change from baseline indicate reduction (improvement) in sino-nasal symptoms.
  units on a scale | 41.5 (20.84)
Nasal Obstruction/Congestion ≥ 2 [Count of Participants; unit: Participants] — Determined on a scale of 0 (no symptoms) to 3 (severe symptoms) based on the subject's recollection of symptoms over the past week using a reflective paper questionnaire. Negative values for change from baseline to follow-up indicate reduction (improvement) in nasal obstruction/congestion.
  Participants | 38
Ethmoid Sinus Obstruction [Mean (Standard Deviation); unit: percent of obstruction] — Estimated visually based on endoscopic examination on a scale of 0% (no obstruction) to 100% (complete obstruction of the ethmoid cavity by polyps, edema, and/or scarring).
  percent of obstruction | 73.2 (22.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Implant-Related Serious Adverse Events
Description: Evaluated via tabulation of implant-related serious adverse events (SAE) reported by subjects between consent and Day 365.
Time Frame: 365 days
Measure: Count of Participants; unit: Participants
Groups:
- S8 Sinus Implant: Corticosteroid-eluting Sinus Implant with 1350 mcg of MF
  Mometasone furoate nasal spray (MFNS, 200 mcg) once daily
Arm/Group | S8 Sinus Implant
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: SNOT-22 Total Score
Description: Sino-Nasal Outcomes Test (SNOT-22) is a validated disease-specific symptom-scoring instrument consisting of 22 questions, each scored on a 6-point scale of 0 (no problem) to 5 (probably as bad as it can be) based on the subject's recollection of symptoms over the past 2 weeks. The total score ranges from 0 to 110, with a higher score reflecting greater symptom burden. Change from baseline to 90 days and to 180 days is calculated as the value at 90/180 days minus the value from baseline. Negative values for change from baseline indicate reduction (improvement) in sino-nasal symptoms.
Time Frame: Baseline, 90 days, 180 days
Population: Analysis population includes subjects with available data at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- S8 Sinus Implant: Corticosteroid-eluting Sinus Implant with 1350 mcg of MF
  MFNS (200 mcg) once daily)
Arm/Group | S8 Sinus Implant
Number analyzed (Participants) | 50
score on a scale
  Change from baseline to Day 90 | -14.9 (19.27)
  Change from baseline to Day 180 | -15.4 (20.36)

3. Secondary Outcome: Nasal Obstruction/Congestion Score
Description: Determined on a scale of 0 (no symptoms) to 3 (severe symptoms) based on the subject's recollection of symptoms over the past week using a reflective paper questionnaire. Change from baseline to 90 days and to 180 days is calculated as the value at 90/180 days minus the value at baseline. Negative values for change from baseline to follow-up indicate reduction (improvement) in nasal obstruction/congestion.
Time Frame: Baseline, 90 days, 180 days
Population: Analysis population includes subjects with available data at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- S8 Sinus Implant: Corticosteroid-eluting Sinus Implant with 1350 mcg of MF.
  MFNS (200 mcg) once daily
Arm/Group | S8 Sinus Implant
Number analyzed (Participants) | 50
units on a scale
  Change from baseline to Day 90 | -0.6 (0.91)
  Change from baseline to Day 180 | -0.6 (0.94)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through Day 365.
Groups:
- S8 Sinus Implant: Corticosteroid-eluting Sinus Implant with1350 mcg MF.
  MFNS (200 mcg) once daily
Arm/Group | S8 Sinus Implant
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S8 Sinus Implant (N=50)
brain hypoxia (Nervous system disorders) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
small intestine obstruction (Gastrointestinal disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S8 Sinus Implant (N=50)
acute sinusitis (Infections and infestations) | 2 (2) — implant-related adverse event
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) — implant-related adverse event
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) — implant-related adverse event
rhinalgia (Respiratory, thoracic and mediastinal disorders) | 3 (3) — implant-related adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03358329/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT03358329/SAP_001.pdf